CLINICAL TRIAL: NCT02047071
Title: Effect of Continuous Positive Airways Pressure (CPAP) in Women With Moderate-to-severe Obstructive Sleep Apnea (OSA). A Multicenter, Randomized, Controlled Trial.
Brief Title: Effect of CPAP Treatment in Women With Moderate-to-severe OSA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Campos-Rodriguez (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor-Investigator, Francisco Campos-Rodriguez, Pneumology specialist, Sociedad Española de Neumología y Cirugía Torácica
Organization: Sociedad Española de Neumología y Cirugía Torácica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI13/00743
Record Dates: First submitted 2014-01-19; First posted 2014-01-28 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Female gender; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Conservative treatment. This group will be receive standard care for OSA consisting of hygienic-dietary advice and lifestyle counseling.
- Continuous positive airways pressure (Experimental): Optimal Continuous positive airways pressure treatment every night plus standard care for OSA consisting of hygienic-dietary advice and lifestyle counseling.
  Interventions: Device: Continuous positive airways pressure

INTERVENTIONS:
Device: Continuous positive airways pressure — Optimal Continuous positive airways pressure treatment every night plus standard care for OSA consisting of hygienic-dietary advice and lifestyle counseling.
  Arms: Continuous positive airways pressure

SUMMARY:
The purpose of this study is to determine whether Continuous Positive Airways Pressure (CPAP) improves quality of life, cardiovascular (blood pressure) and metabolic profile (glucose and lipid metabolism) in females with moderate-to-severe Obstructive Sleep Apnea (OSA).

DETAILED DESCRIPTION:
Study Design: multicenter, open-label, randomized, controlled trial of parallel groups with a final blind evaluation.

Study sites. The following hospitals will participate in the study: Valme (Sevilla), la Fe (Valencia), Virgen del Rocío (Sevilla), Gral Yagüe (Burgos), San Pedro de Alcántara (Cáceres), Dr Peset (Valencia), Severo Ochoa (Madrid), Reina Sofía (Córdoba), Dr Negrín (Las Palmas de Gran Canaria), Virgen de la Victoria (Málaga), Río Hortega (Valladolid), Costa del Sol (Málaga), Marqués de Valdecilla (Santander), Albacete (Albacete), Virgen del Puerto (Cáceres), Puerta de Hierro (Madrid), Consorcio Sanitario de Terrassa (Barcelona), Getafe (Madrid), Gral de Alicante (Alicante), Morales Meseguer (Murcia), Tomelloso (Ciudad Real), and Fundación Jiménez Díaz (Madrid). All centers from Spain.

Methods: consecutive outpatient women aged 18-75 years and referred to the sleep clinics for suspicion of OSA will be studied. They will undergo a diagnostic home respiratory polygraphy, and those diagnosed with moderate-to-severe OSA (AHI ≥15) will be eligible for this study and randomized to optimal CPAP treatment or conservative treatment for 12 weeks. Every women will fulfill a standardized protocol and different quality of life questionnaires. Office blood pressure will be measured. Fasting blood samples will be collected to assess glucose and lipid metabolism. All the measurements will be performed at baseline and after 12 weeks of follow-up. Women will be examined at the time of inclusion, after 4 weeks of follow-up and at the end of follow-up (12 weeks).

149 women with moderate-to-severe OSA need to be enrolled in each study arm, according to the sample size calculated to achieve a clinically significant improvement in the Quebec Sleep Questionnaire. The results will be analyzed both on an intention-to-treat basis and on a per-protocol basis (data only from patients who finish the study and show good adherence to CPAP, defined as an average objective use of at least 4 hours/day).

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe OSA (Apnea-Hypopnea index ≥15) diagnosed by Home Respiratory Polygraphy.
* Age between 18-75 years.

Exclusion Criteria:

* diagnosis of narcolepsy or restless legs syndrome
* unstable cardiovascular profile (cardiovascular event in the previous 3 months)
* cancer or life expectancy lower than 1 year
* uncontrolled psychiatric disorders
* central sleep apnea (>50% of central events)
* pregnancy
* risky jobs and severe hypersomnolence (Epworth >=18) requiring urgent treatment
* either respiratory failure (SaO2<90% or partial oxygen pressure [pO2] <60 mmHg or Long-term O2 therapy
* heart failure (New York Heart Association class III-IV)
* prior CPAP therapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2014-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of life on the Quebec Sleep Questionnaire (QSQ) at week 12 | Baseline, 12 weeks.

SECONDARY OUTCOMES:
Change from baseline in quality of life on the 12-Item Short Form Health Survey (SF-12) at week 12 | baseline, 12 weeks
Change from baseline in mood state on the Abbreviated Profile Of Mood States (POMS) at week 12 | Baseline, 12 weeks
Change from baseline in sleepiness on the Epworth Sleepiness Score (ESS) at week 12 | baseline, 12 weeks
Change from baseline in anxiety and depression on the Hospital Anxiety and Depression questionnaire (HAD) at week 12 | baseline, 12 weeks
Change from baseline in quality of life on the Visual Analogic Scale (VAS) at week 12 | baseline, 12 weeks
Change from baseline in sleep apnea symptoms at week 12 | baseline, 12 weeks
Change from baseline in blood pressure at week 12 | Baseline, 12 weeks
  Change in office blood pressure from baseline at week 12
Change from baseline in glucose metabolism at week 12 | baseline, 12 weeks
Change from baseline in lipid metabolism at week 12 | baseline, 12 weeks

OTHER OUTCOMES:
Number of Participants with CPAP use >= 4 hours/day as a Measure of CPAP adherence | Baseline, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Campos-Rodriguez, MD, Principal Investigator — Sociedad Española de Neumología y Cirugía Torácica
Locations (1):
- Hospital Universitario Valme, Seville, Spain

REFERENCES:
- [Derived] Campos-Rodriguez F, Asensio-Cruz MI, Cordero-Guevara J, Jurado-Gamez B, Carmona-Bernal C, Gonzalez-Martinez M, Troncoso MF, Sanchez-Lopez V, Arellano-Orden E, Garcia-Sanchez MI, Martinez-Garcia MA; Spanish Sleep Network. Effect of continuous positive airway pressure on inflammatory, antioxidant, and depression biomarkers in women with obstructive sleep apnea: a randomized controlled trial. Sleep. 2019 Oct 9;42(10):zsz145. doi: 10.1093/sleep/zsz145. PMID 31314107
- [Derived] Campos-Rodriguez F, Gonzalez-Martinez M, Sanchez-Armengol A, Jurado-Gamez B, Cordero-Guevara J, Reyes-Nunez N, Troncoso MF, Abad-Fernandez A, Teran-Santos J, Caballero-Rodriguez J, Martin-Romero M, Encabo-Motino A, Sacristan-Bou L, Navarro-Esteva J, Somoza-Gonzalez M, Masa JF, Sanchez-Quiroga MA, Jara-Chinarro B, Orosa-Bertol B, Martinez-Garcia MA; Spanish Sleep Network. Effect of continuous positive airway pressure on blood pressure and metabolic profile in women with sleep apnoea. Eur Respir J. 2017 Aug 10;50(2):1700257. doi: 10.1183/13993003.00257-2017. Print 2017 Aug. PMID 28798089
- [Derived] Campos-Rodriguez F, Queipo-Corona C, Carmona-Bernal C, Jurado-Gamez B, Cordero-Guevara J, Reyes-Nunez N, Troncoso-Acevedo F, Abad-Fernandez A, Teran-Santos J, Caballero-Rodriguez J, Martin-Romero M, Encabo-Motino A, Sacristan-Bou L, Navarro-Esteva J, Somoza-Gonzalez M, Masa JF, Sanchez-Quiroga MA, Jara-Chinarro B, Orosa-Bertol B, Martinez-Garcia MA; Spanish Sleep Network. Continuous Positive Airway Pressure Improves Quality of Life in Women with Obstructive Sleep Apnea. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Nov 15;194(10):1286-1294. doi: 10.1164/rccm.201602-0265OC. PMID 27181196